CLINICAL TRIAL: NCT00003733
Title: A Phase II Study of Sequential Carboplatin, Paclitaxel and Hycamtin in Patients With Previously Untreated Advanced Ovarian Cancer
Brief Title: Sequential Chemotherapy in Treating Patients With Residual Disease Following Surgery for Stage IIB, Stage III, or Stage IV Ovarian Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: SmithKline Beecham (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066848; SB-104864/289; EU-98068
Record Dates: First submitted 1999-11-01; First posted 2004-06-09 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2000-12

CONDITIONS: Ovarian Cancer
Keywords: stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Carboplatin; Paclitaxel; Topotecan

INTERVENTIONS:
Drug: carboplatin
Drug: paclitaxel
Drug: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving chemotherapy drugs in different ways may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of sequential chemotherapy in treating patients with residual disease following surgery for stage IIB, stage III, or stage IV ovarian cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the efficacy of sequential carboplatin, paclitaxel, and topotecan in terms of disease response, time to progression, survival and progression free survival in patients with stage IIB, stage III, or stage IV ovarian epithelial cancer. II. Assess the toxicity of this regimen in this patient population.

OUTLINE: Patients receive carboplatin IV over 30 to 60 minutes on days 1 and 22. Patients then receive paclitaxel IV over 3 hours on days 43 and 64, then topotecan IV over 30 minutes daily for 5 days beginning on days 85, 106, 127, and 148. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients are followed monthly for 3 months and then every 3 months for 2 years.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed advanced ovarian epithelial carcinoma with greater than 1 cm residual disease at completion of initial surgery Stage IIB, IIIA, IIIB, IIIC, or IV Measurable disease OR CA 125 greater than 120 units/mL obtained post surgery

PATIENT CHARACTERISTICS: See General Eligibility Criteria

PRIOR CONCURRENT THERAPY: Biological therapy: No prior or concurrent immunotherapy Chemotherapy: No prior or concurrent chemotherapy Endocrine: No prior or concurrent hormonal therapy Radiotherapy: No prior radiotherapy No concurrent radiotherapy except to limited fields (e.g., for palliation of bone pain) Surgery: Diagnostic surgery performed less than 12 weeks prior to study No concurrent interval debulking Other: At least 30 days or five half-lives since any prior investigational therapy No other concurrent investigational therapy --Patients Characteristics-- Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Hemoglobin at least 9.0 g/dL WBC at least 4,000/mm3 Neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: SGOT and/or SGPT no greater than 2.5 times upper limit of normal (ULN) (no greater than 5 times ULN if liver metastases present) Alkaline phosphatase no greater than 2.5 times ULN (no greater than 5 times ULN if liver and/or bone metastases present) Renal: Creatine less than 2 times ULN Creatinine clearance at least 50 mL/min Other: No prior malignancy except basal cell skin carcinoma or carcinoma in situ of the cervix No uncontrolled infection No other concurrent medical conditions that would prevent full compliance or expose patient to extreme risk or decreased life expectancy No concurrent medical condition for which treament with platinum compounds is contraindicated No history of allergy to compounds related to the drugs used in this study No prior motor or sensory neurotoxicity grade 2 or worse Not pregnant or nursing Fertile patients must use effective contraception

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 1997-12

CONTACTS AND LOCATIONS:
Overall Officials: Gordon J.S. Rustin, MD, Study Chair — Mount Vernon Cancer Centre at Mount Vernon Hospital
Locations (2):
- United Kingdom (2):
  - Charing Cross Hospital, London, England
  - Mount Vernon Hospital, Northwood, England

REFERENCES:
- [Result] Guppy AE, Nelstrop AE, Foster T, Agarwal R, Seckl MJ, Rustin GJ. A phase II study of sequential carboplatin, paclitaxel and topotecan in patients with previously untreated advanced ovarian cancer. Br J Cancer. 2004 Feb 23;90(4):810-4. doi: 10.1038/sj.bjc.6601618. PMID 14970858